CLINICAL TRIAL: NCT04721886
Title: Interstitial Fluid Pressure Estimation in Breast Cancer Using 3D Subharmonic Signals From Contrast-Enhanced Ultrasound
Brief Title: Contrast-Enhanced Ultrasound Scan for the Estimation of Tissue Pressure in Patients With Breast Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20G.605
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves; perflutren

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (CEUS) (Experimental): Patients undergo ultrasound without contrast. Patients then receive Definity IV over 15 minutes and undergo CEUS.
  Interventions: Procedure: Ultrasonsgraphy; Drug: Perflutren Lipid Microcpheres; Procedure: Contrast - Enhanced Ultrasound

INTERVENTIONS:
Procedure: Ultrasonsgraphy — Undergo ultrasonography
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; ultrasound; Ultrasound Imaging; Ultrasound Test; Medical; US
Drug: Perflutren Lipid Microcpheres — Given IV
  Other Names: Definity
Procedure: Contrast - Enhanced Ultrasound — Undergo CEUS
  Other Names: CEUS

SUMMARY:
This clinical trial studies the use of contrast-enhanced ultrasound (CEUS) in estimating tissue pressure in patients with breast cancer. Diagnostic procedures, such as CEUS, may help estimate tissue pressure noninvasively.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the 3-dimensional (3D) subharmonic aided pressure estimation (SHAPE) results can be used to estimate interstitial fluid pressures (IFPs) in breast tumor and its surrounding tissue.

SECONDARY OBJECTIVE:

I. To determine if the malignancy of breast tumor can be predicted by the 3D SHAPE results.

OUTLINE:

Patients undergo ultrasound without contrast. Patients then receive perflutren lipid microspheres (Definity) intravenously (IV) over 15 minutes and undergo CEUS.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Be conscious, willing and able to comply with all study procedures and be available for the duration of the study
* At least 21 years old
* Be scheduled for a breast biopsy (Breast Imaging Reporting and Data System [BIRAD] 4, 4A, 4B, 4C or 5)
* Patient with an at least 1 cm mass located at < 3 cm depth, approachable by 2.5 inch needle
* Be medically stable as determined by the investigator
* If a female of child-bearing potential, must have a negative urine pregnancy test within 24 hours prior to administration of Definity

Exclusion Criteria:

* Females who are pregnant or nursing
* Patients who are medically unstable, patients who are seriously or terminally ill, and patients whose clinical course is unpredictable. For example:
* Patients on life support or in a critical care unit
* Patients with unstable occlusive disease (e.g., crescendo angina)
* Patients with clinically unstable cardiac arrhythmias, such as recurrent ventricular tachycardia
* Patients with uncontrolled congestive heart failure (New York Heart Association [NYHA] class IV)
* Patients with recent cerebral hemorrhage
* Patients who have undergone surgery within 24 hours prior to the study sonographic examination
* Patients with known hypersensitivity or allergy to any component of Definity
* Patients with unstable cardiopulmonary conditions or respiratory distress syndrome
* Patients with uncontrollable emphysema, pulmonary vasculitis, pulmonary hypertension or a history of pulmonary emboli

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between subharmonic aided pressure estimation (SHAPE) results and direct measurements of interstitial fluid pressure (IFP) | At baseline
  Pearson's correlation coefficients will be computed between SHAPE results and direct IFP measurements by Stryker compartment pressure monitoring system. A Pearson's correlation coefficient above 0.5 will be considered a successful outcome.

SECONDARY OUTCOMES:
Prediction of malignancy of breast tumor by the 3-dimensional subharmonic aided pressure estimation results | At baseline
  Generalized linear mixed logistic or generalized estimating equations logistic modeling of tumor versus non-tumor samples will be used to explore the potential for using SHAPE results as a novel functional predictor of breast tumor malignancy. Additionally, the subharmonic signal ratio from the tumor will be used to predict the malignancy of breast tumor using a biopsy result as a gold standard. The Mann-Whitney or Student's t-test will be performed depending on the distribution of the results.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States